CLINICAL TRIAL: NCT06933485
Title: Posture-Focused Exercise Program for Dental Students: A Preliminary Evaluation
Brief Title: Posture and Prevention: Evaluating an Exercise Program for Dental Students
Acronym: Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Alime Buyuk, Principal Investigator, PhD., Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6553; TÖBAP-2024-6553 (Other Grant/Funding Number: Akdeniz University)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Postural Instability; Dentistry; Musculoskeletal
Keywords: postural disorders; dentistry students; pain; exercises; musculoskeletal disease
MeSH Terms: conditions — Pain; Motor Activity; Musculoskeletal Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postural exercise group (Experimental): The intervention group contains a combination of the postural exercises and education. One hour of each training consists of the postural exercise practice and education
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — These sessions of the postural exercise aim to increase student's knowledge and awarenes their benefits for trunk stabilization, posture correction and diaphragmatic breathing will be explained by the expert physiotherapist. In the exercise planning; the exercise session start with warm-up exercises; A transition to the flow of exercise is ensured with warm-ups that include arm, leg and trunk movements for approximately 10 minutes, and then all extremities are worked for approximately 40 minutes in the main exercise session to ensure trunk alignment. The last 10 minutes of the exercise session is completed with approximately 10 minutes of cool-down exercises to which light stretching is added, making the exercise session a total of 60 minutes.

SUMMARY:
Musculoskeletal disorders (MSDs) are a major public health concern, involving inflammatory and degenerative issues in muscles, tendons, joints, and nerves. Commonly caused by repetitive strain and poor posture, these disorders are highly prevalent among dental professionals due to their physically demanding work environments.

Studies show that 64% to 93% of dentists experience MSDs during their careers, often beginning during dental education. Dental students, exposed to hands-on clinical training from early on, face physical strain without sufficient ergonomic awareness. Poor working posture, prolonged procedures, and static positions increase the risk significantly.

Recent findings at Akdeniz University reveal that 90.8% of fourth- and fifth-year dental interns reported MSD symptoms, especially in the neck, back, and shoulders. Alarmingly, only 21.7% engaged in regular physical activity, although 85.5% were interested in learning preventive exercises.

These results underline the urgent need for early ergonomic education and physical activity. Even with proper posture, over 50% of muscles remain contracted to maintain dental working positions, leading to fatigue and pain. Incorporating structured, posture-oriented stretching and strengthening exercises can help prevent these issues.

Scientific studies confirm that regular stretching improves joint lubrication, circulation, and muscular relaxation, while reducing pain and preventing trigger points. Short sessions during clinical work have been shown to reduce MSD symptoms effectively.

In response, a Posture-Oriented Exercise Program is being developed for Akdeniz University dental students under physiotherapy guidance. Supported by the Özlenen Student Scientific Research Project, this initiative aims to raise awareness, promote musculoskeletal health, and build long-term professional well-being. The program includes practical, supervised exercises and will evaluate outcomes such as posture, pain levels, and ergonomic habits.

This project could serve as a model for integrating physical health education into dental curriculums, improving both student welfare and the sustainability of dental practice.

DETAILED DESCRIPTION:
Musculoskeletal disorders (MSDs), which are increasingly common worldwide and defined as a significant public health problem, include inflammatory and degenerative conditions affecting muscles, tendons, ligaments, nerves, bones, and joints. These problems, which mainly develop due to cumulative trauma from repetitive-strain movements and ergonomic deficiencies, negatively affect individuals' daily living activities by causing pain, restricted movement, and injuries.

Due to the limited working area of the oral cavity and long working hours, dentists are a high-risk group for MSDs. Working in a bent and overly strained posture during dental procedures, keeping the arm in fixed positions for long periods, making repetitive and usually forceful movements, sitting or standing for extended periods, using high-vibration tools, and being exposed to various psychosocial stressors all play a significant role in the development of MSDs in dentists. Literature shows that between 64% and 93% of dentists experience MSDs at some point in their careers. While these are common health problems, they can decrease healthcare workers' productivity, lead to high economic costs, and negatively affect individuals' quality of life.

Musculoskeletal disorders can begin during dental school and continue throughout professional life if preventive and corrective measures are not taken. Unlike other disciplines, dental education includes both theoretical and clinical training concurrently over five years. Students practice hand-eye coordination-based applications during the first three years through preclinical education alongside theoretical courses. In the final two years, they begin physically demanding clinical internships. At this stage, without sufficient clinical experience and ergonomic awareness, students may ignore physical warning signs to gain a better field of view, leading to improper repetitive movements and maintaining abnormal or static postures for extended durations.

Even in ideal working positions, dentists must contract over 50% of their muscles to maintain a stable posture against gravity. Any deviation from the spine's natural four curves - cervical lordosis, thoracic kyphosis, lumbar lordosis, and sacral kyphosis - places extra stress on muscles, ligaments, or soft tissue to keep the spine upright. These postures lead to prolonged, repetitive muscle contractions typical among dentists, causing muscle imbalances. Incorrect posture accelerates degeneration in vertebrae, discs, muscles, and ligaments, leading to pain.

Research from various countries has shown that MSD symptoms can begin during dental education. For example, a study on Australian dental students found that 84.6% had MSDs caused by clinical internships. The same study revealed that 61% of students had incorrect posture. Therefore, it's crucial to raise awareness about the prevalence of MSDs and ergonomic principles starting from dental school years.

In 2022, as part of the "Ergonomics and Stretching Movements in Dentistry" course within the Special Study Module of the Department of Periodontology, a study with third-year students has been made in Akdeniz University. Among the fourth- and fifth-year dental interns who participated, 90.8% reported musculoskeletal complaints in at least one body region over the past 12 months. The most frequently affected areas were the neck (80.9%), back (71.7%), lower back (69.1%), and shoulders (65%). Additionally, 14.5% had visited a doctor due to pain, 9.2% had taken leave or received a medical report, and 4% had used medication. Alarmingly, only 21.7% of the participants reported engaging in regular physical activity, and nearly all (85.5%) expressed a desire for training on preventive stretching and exercises in dentistry.

By nature, the human body needs to move. Yet, technological advancements have led people toward sedentary lifestyles, which are incompatible with human physiology and increase the risk of disease. Regular and conscious physical activity not only promotes a healthy body structure but also releases hormones that make individuals more energetic, happier, and psychologically balanced. For a healthier society, the habit of daily physical activity should be taught from a young age as an indispensable part of life. Unfortunately, the increasingly demanding theoretical and clinical training in dentistry leaves students with little time for hobbies. Similar studies in other countries have also reported that dental students struggle to maintain regular exercise routines. As a result, dentists are now among the professionals who increasingly seek physical therapy and ergonomic advice.

Recent studies have shown growing interest in regular exercise programs to reduce work-related MSD risk among dentists. Stretching exercises are known to improve blood circulation, increase synovial fluid for joint lubrication, reduce painful trigger points, and help relax muscles. These benefits can significantly impact both the personal and professional lives of dentists. Research indicates that stretching exercises performed during periodic chairside breaks can reduce MSD-related complaints. A randomized controlled study showed that six weeks of neck exercises in women with chronic neck pain significantly improved cervical angles and posture, as observed via imaging systems. Similarly, a 10-week neck and shoulder exercise program positively affected the working posture of dental students.

Considering all of this, this study believed that raising awareness among young dental students about the importance of regular physical activity can help prevent future MSDs. For this purpose, in this study - supported by the Özlenen Student Scientific Research Project and designed as a social responsibility initiative - aims to implement a posture-focused exercise program for dental students at Akdeniz University Faculty of Dentistry, guided by an experienced physiotherapist, and evaluate the outcomes of these physical activities.

ELIGIBILITY:
Inclusion Criteria:

* Being a student studying at Akdeniz University Faculty of Dentistry
* Individuals who volunteer to participate in the study
* No harm to exercise by the doctor
* Participants who experienced musculoskeletal pain during the past 3 month, at least in one of the examined body regions (i.e., the neck, shoulders, upper back and lower back)

Exclusion Criteria:

* History of traumatic or surgical intervention of spine
* Any orthopedic, neurological, respiratory, or circulatory disorders
* Participation in professional sports training or a structured exercise program within the previous six months
* The current use of pain medications or muscle relaxants.
* Being over 25 years

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Quality Of Life Questionnaire | 1 week
  The study uses the Short-Form-36 (SF-36) questionnaire to collect information about the participant's health-related quality of life (QOL). The SF-36 assesses eight domains of health-related QOL, namely, physical functioning (PF), role limitations due to physical problems (RP), role limitations due to emotional problems (RE), energy/vitality (V), mental health (MH), social functioning (SF), bodily pain (BP), and general perception of health (GH). Each dimension is scored from 0 to 100 %, with higher scores indicating a better quality of life. In this study, both the eight subscale scores and the two summary measures including the physical component summary (PCS) (a sum of scores of functional capacity, physical aspects, pain, and general health divided into 4) and the mental component summary (MCS) (a sum of vitality, social aspects, emotional aspects, and mental health divided into 4) were evaluated.
Nordic Musculoskeletal Questionnaire (NMQ-7) | 1 week
  The modified NORDIC questionnaire questions whether there is pain on a figure that anatomically shows nine areas of the body (neck, shoulder, back, elbow, hand/wrist, waist, hip/thigh, knee, foot/ankle) and the severity of this pain (0 points no pain, 10 points the most severe pain known) with the Visual Analog Scale (VAS).
Spinal Mobility | 1 week
  Spinal Mouse Device: Thoracic angle and lateral inclination of the spine measures with the Spinal Mouse device (Idiag, Fehraltorf, Switzerland), which is a non-invasive, computer-aided, easy-to-use device that provides valid and reliable results when compared to radiographic analyses. The measurements are maden by a physiotherapist. The patient's demographic information (name, surname, gender, year of birth) is recorded on the computer with the Spinal Mouse device software. The patient is asked to stand in the most comfortable position with their back visible. The Spinal Mouse device is placed on the 7th cervical vertebra and the recording is started by pressing the button on it. The device moves on the skin from the 7th cervical vertebra to the 3rd sacral vertebra along the line of the spinous processes marked by its wheels. After reaching the sacral 3 level, the recording is completed by pressing the button on the device again.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Kustarcı, Profesor, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University Destistry Faculty, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It's written by Turkish language